CLINICAL TRIAL: NCT04339244
Title: Effect of Arterial Pressure Regulation on Optic Nerve Sheath Diameter During Robot Assisted Laparoscopic Surgery
Brief Title: Effect of Pressure Regulation on Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Principal Investigator, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-07-049
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: arterial pressure regulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONSD measurement under lower blood pressure (Active Comparator): ONSD measurement under mean blood pressure of 60~70 mmHg
  Interventions: Other: RALRP under lower mean BP
- ONSD measurement under highly normal blood pressure (Active Comparator): ONSD measurement under mean blood pressure of 90~100 mmHg
  Interventions: Other: RALRP under lower mean BP

INTERVENTIONS:
Other: RALRP under lower mean BP — RALRP under regulation of lower mean BP
  Arms: ONSD measurement under lower blood pressure
Other: RALRP under lower mean BP — RALRP under regulation of highly normal mean BP
  Arms: ONSD measurement under highly normal blood pressure

SUMMARY:
Intracranial pressure is known to increase during robot-assisted laparoscopic radical prostatectomy (RALRP) due to steep trendelenberg position. Measurement of optic nerve sheath diameter (ONSD) is a indirect method which can assess the degree of intracranial pressure.

This study is designed to measure the ONSD during RALRP under regulation of arterial pressure.

DETAILED DESCRIPTION:
During last decades, RALRP has been advocated due to the advantages of short hospital stay, reduced blood loss during surgery, less postoperative pain and complication. During RALRP, steep trendelenberg postion and pneumoperitoneum are required essentially, and this is for the acquisition of adequite surgical field. However, such position and pneumoperitoneum can result in harmful hemodynamic change. Previous study demonstrated that patients of RALRP showed 12.5% increase of ONSD.

The relationship of ONSD and increase of intracranial pressure has been proved previously through many studies. Recent meta analysis showed that ONSD measurement for the monitor of ICP demonstrated that sensitivity 0.9, specificity 0.85 and ROC cuve 0.983.

In addition, increase of ONSD during RALRP can be affected by the degree of arterial pressure and end tidal CO2 increase.

This study is designed to see the effect of arterial pressure regulation on the increase of ONSD

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer receiving RALRP

Exclusion Criteria:

* glaucoma
* intracranial tumor
* previous disease elevating intracranial pressure

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath diameter change among 4 time period | Baseline, 1 hour, 2 hours, 2.5 hours after completion of the intervention
  optice nerve sheath diameter change among 4 time period

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Jung, PhD, Study Director — 82532584892
Locations (1):
- Hong ji HEE, Daegu, South Korea